CLINICAL TRIAL: NCT03633799
Title: A Phase 3, Prospective, Multi-Center, Single-Arm, Open-Label Study to Evaluate VeraCept®, a Long-Acting Reversible Intrauterine Contraceptive for Contraceptive Efficacy, Safety, and Tolerability
Brief Title: Evaluation of Efficacy, Safety and Tolerability of VeraCept IUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sebela Women's Health Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Organization: Sebela Pharmaceuticals Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMDOC-0042
Record Dates: First submitted 2018-07-19; First posted 2018-08-16 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Women at Risk for Pregnancy

STUDY DESIGN:
Intervention Model Description: VeraCept Intrauterine System (IUS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VeraCept (Experimental): VeraCept® Intrauterine Contraceptive
  Interventions: Drug: VeraCept

INTERVENTIONS:
Drug: VeraCept — VeraCept Intrauterine Contraceptive is a hormone free, low dose, copper-releasing birth control method

SUMMARY:
To assess the contraceptive efficacy (prevention of pregnancy) of VeraCept

DETAILED DESCRIPTION:
Study Design:

Prospective, multi-center, single-arm, open-label, Phase 3 clinical study to 3 years with extension up to 8 years

Number of Subjects:

Approximately 1,605 subjects will be enrolled into the study

Study Population:

Post-menarcheal, pre-menopausal women up to age 45 years, who are at risk for pregnancy and who desire a long-term intrauterine contraceptive for birth control will be eligible for this study.

Primary Endpoint:

The primary endpoint is the contraceptive efficacy through 3 years of use, as assessed by the Pearl Index.

Secondary endpoints:

Contraceptive Efficacy:

* Pearl Index at Years 4, 5, 6, 7 and 8 as well as cumulatively through Years 4, 5, 6, 7 and 8.
* Pregnancy percentage by life table analysis (Kaplan-Meier) at Years 1, 2, 3, 4, 5, 6, 7 and 8
* The cumulative Pearl Index for Years 6 to 8 will be calculated as well as the cumulative pregnancy percentage for Years 6 to 8 using a life table analysis (Kaplan-Meier) only for the EP population.

Study drug placement:

* Ease of VeraCept placement
* Placement success

Safety:

* Serious adverse events (SAEs)
* Adverse events (AEs)
* Pelvic infection (pelvic inflammatory disease (PID) or endometritis)
* Ectopic pregnancies
* Uterine perforations
* Dysmenorrhea
* Abdominal pain
* Expulsion rates at Years 1, 2, 3, 4, 5, 6, 7 and 8

Tolerability:

* Bleeding and spotting patterns
* Insertion pain assessed immediately after insertion
* Continuation rates at Years 1, 2, 3, 4, 5, 6, 7 and 8
* Reasons for discontinuation

Return to fertility

● Pregnancy rate in subjects who request VeraCept removal specifically to become pregnant. Subjects who desire pregnancy after having VeraCept removed will be followed for either 1 year, until they decide to no longer try to conceive or they become pregnant, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menarcheal, pre-menopausal females up to 45 years of age at the time of informed consent/assent and in good general health;
2. History of regular menstrual cycles defined as occurring every 21-35 days when not using hormones or prior to recent pregnancy or spontaneous or induced abortion;
3. Sexually active with a male partner who has not had a vasectomy;
4. Reasonably expect to have coitus at least once monthly during the study period;
5. In a mutually monogamous relationship of at least 3 months duration;
6. Seeking to avoid pregnancy for the duration of the study;
7. Willing to use the study drug as the sole form of contraception;
8. Willing to accept a risk of pregnancy;
9. Subjects must be in compliance with cervical cancer screening guidelines per the American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines without evidence of disease. Subjects who are age 21-24 y/o, at time of informed consent, must have a normal Papanicolaou test (Pap), atypical squamous cells of undetermined significance (ASC-US), or low-grade squamous intraepithelial lesion (LSIL). Subjects who are 25 or older at the time of informed consent with ASC-US results, must also have a negative high-risk human papilloma virus (HPV) test result within the appropriate screen timeframe per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines, and prior to the study IUS insertion. Alternatively, the subject must have had a colposcopy performed within the appropriate screen timeframe, and prior to the study IUS insertion that showed no evidence of dysplasia requiring treatment per ASCCP guidelines, or treatment was performed and follow-up at least 6 months after the treatment showed no evidence of disease by clinical evaluation;
10. Able and willing to comply with all study tests, procedures, assessment tools (including e-diary) and follow-up;
11. Able and willing to provide and document informed consent and Authorization for Release of Protected Health Information (PHI). Unemancipated subjects under 18 years old must provide assent and have written parental consent documented on the consent form consistent with local legal requirements;
12. Plan to reside within a reasonable driving distance of a research site for the duration of the study.
13. Subject agrees not to self-remove VeraCept

Exclusion Criteria:

1. Known or suspected pregnancy; or at risk for pregnancy from unprotected intercourse earlier in current cycle;
2. Subject who anticipates separation from her partner for more than a 6-month period during use of VeraCept;
3. A previously inserted intrauterine system (IUS) that has not been removed by the time the study IUS is placed;
4. History of previous IUS complications, such as perforation, expulsion, or pregnancy with IUS in place;
5. Pain with current IUS;
6. Injection of hormonal contraceptive (e.g., Depo-Provera) within the last 10 months and has not had 2 normal menstrual cycles since the last injection;
7. Planned use of any non-contraceptive estrogen, progesterone or testosterone any time during study participation;
8. Exclusively breastfeeding before return of menses; lactating women will be excluded unless they have had 2 normal menstrual periods prior to enrollment;
9. Unexplained abnormal uterine bleeding (suspicious for a serious condition), including bleeding 4 weeks post-septic abortion or puerperal sepsis;
10. Severely heavy or painful menstrual bleeding;
11. Suspected or known cervical, uterine or ovarian cancer, or unresolved clinically significant abnormal Pap smear requiring evaluation or treatment;
12. Any history of gestational trophoblastic disease with or without detectable elevated ß-human chorionic gonadotropin (ß-hCG) levels, or related malignant disease;
13. Any congenital or acquired uterine anomaly that may complicate study drug placement, such as:

    * Submucosal uterine leiomyoma
    * Asherman's syndromes
    * Pedunculated polyps
    * Bicornuate uterus
    * Didelphus or uterine septa
14. Any distortions of the uterine cavity (e.g. fibroids), that, in the opinion of the investigator, are likely to cause issues during insertion, retention or removal of the IUS;
15. Known anatomical abnormalities of the cervix such as severe cervical stenosis, prior trachelectomy or extensive conization that, in the opinion of the investigator would prevent cervical dilation and study drug placement;
16. Untreated or unresolved acute cervicitis or vaginitis;
17. Known or suspected human immunodeficiency virus (HIV) infection or clinical AIDS;
18. Subjects who have an established immunodeficiency;
19. Known intolerance or allergy to any components of VeraCept including intolerance or allergy to nickel, titanium, or copper, and including Wilson's Disease;
20. Currently participating or planning future participation in a research study of an investigational drug or device during the course of this investigational study. Subject must have waited at least 30 days from exiting their last study prior to informed consent in this study;
21. Subject has been enrolled in a previous VeraCept or LevoCept study; 21a. Subject has been enrolled in a previous VeraCept or LevoCept study where VeraCept or LevoCept placement was successful or attempted (replaces exclusion #21 for PK sub-study subjects only);
22. Known or suspected alcohol or drug abuse within 12 months prior to the screening visit;
23. Any general health, mental health or behavioral condition that, in the opinion of the investigator, could represent an increased risk for the subject or would render the subject less likely to provide the needed study information;
24. Study staff or a member of the immediate family of study staff.
25. Subject is <4 weeks post-pregnancy (postpartum, spontaneous or induced abortion)

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only women who are at risk for pregnancy will be eligible for this study
Enrollment: 1620 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2027-09-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, MPH, Principal Investigator — University of Utah
Locations (41):
- United States (41):
  - MomDoc Women's Health Research, Scottsdale, Arizona
  - Copperstate OB/GYN Associates, Tucson, Arizona
  - Essential Access Health, Berkeley, California
  - Essential Access Health, Los Angeles, California
  - Empire Clinical Research, Pomona, California
  - University of California, Davis Health System, Sacramento, California
  - M3 Wake Research (formerly Women's Health Care Research), San Diego, California
  - M3 Wake Research (formerly Medical Center for Clinical Research), San Diego, California
  - Stanford University, Medical Center, Obstetrics and Gynecolocy, Stanford, California
  - Velocity Clinical Research (formerly Downtown Women's Health Care), Englewood, Colorado
  - Altus Research, Inc, Lake Worth, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Women's Health Advantage, Fort Wayne, Indiana
  - Indiana University, Indianapolis, Indiana
  - Praetorian Pharmaceutical Research, Marrero, Louisiana
  - University of Michigan Von Voigtlander Women's Hospital, Ann Arbor, Michigan
  - Planned Parenthood North Central States - Minneapolis, Minneapolis, Minnesota
  - Planned Parenthood Great Rivers (formerly Planned Parenthood of the St. Louis Region and Southwest Missouri), Manchester, Missouri
  - Rex Garn Mabey Jr., MD, Las Vegas, Nevada
  - Capital Health Lawrence OBGYN Research (formerly Lawrence OB/Gyn Clinical Research), Lawrenceville, New Jersey
  - Columbia University Medical Center, Division of Family Planning, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati/Reproductive Medicine Research, Cincinnati, Ohio
  - The Ohio State University Ob/Gyn Research Office, Columbus, Ohio
  - OHSU Women's Health Research Unit, Portland, Oregon
  - University of Pennsylvania/Penn Family Planning and Pregnancy Loss Center, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Center for Family Planning Research, Pittsburgh, Pennsylvania
  - Medical Research South, LLC, Charleston, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Advanced Research Associates, Corpus Christi, Texas
  - Advances In Health, Pearland, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - University of Utah Healthcare Health Sciences Center, Salt Lake City, Utah
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Eastern Virginia Medical, Norfolk, Virginia
  - Seattle Clinical REsearch Center (formerly Seattle Women's Health), Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Creinin MD, Gawron LM, Roe AH, Blumenthal PD, Boraas CM, Hou MY, McNicholas C, Schreifels MJ, Peters K, Culwell K, Turok DK; Copper 175mm(2) IUD Phase 3 Clinical Investigator Group. Three-year efficacy, safety, and tolerability outcomes from a phase 3 study of a low-dose copper intrauterine device. Contraception. 2025 Mar;143:110771. doi: 10.1016/j.contraception.2024.110771. Epub 2024 Nov 22. PMID 39581486

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VeraCept
Started | 1620
Completed | 689
Not Completed | 931
Not completed — Adverse Event | 349
Not completed — Withdrawal by Subject | 288
Not completed — Lost to Follow-up | 97
Not completed — Physician Decision | 9
Not completed — Protocol Violation | 4
Not completed — Pregnancy | 20
Not completed — other | 39
Not completed — ongoing within third year of study | 106
Not completed — unsuccessful study drug placement | 19

BASELINE CHARACTERISTICS:
Arm/Group | VeraCept
Number analyzed (Participants) | 1620
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1620
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 308
  Not Hispanic or Latino | 1312
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18
  Asian | 86
  Native Hawaiian or Other Pacific Islander | 10
  Black or African American | 238
  White | 1196
  More than one race | 62
  Unknown or Not Reported | 10

OUTCOME MEASURES:

1. Primary Outcome: Contraceptive Efficacy Through 3 Years of Use
Description: Contraceptive efficacy through 3 years of use, as assessed by the Pearl Index. The Pearl Index is calculated as the number of on-treatment pregnancies per 100 woman-years of exposure. On-treatment pregnancy is defined as the estimated conception date being on or after the insertion date (must be a successful insertion) and no more than 7 days after the study drug is removed or expelled. One women year is defined as comprising thirteen 28-day cycles. A lower Pearl Index indicates greater contraceptive effectiveness.
Time Frame: 3 years
Population: Evaluable for pregnancy population
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | VeraCept
Number analyzed (Participants) | 1397
Pearl Index | 1.06 [0.67 to 1.61]

2. Secondary Outcome: Contraceptive Efficacy at Years 4, 5, 6, 7 and 8
Description: Pearl Index will be calculated for Years 4, 5, 6, 7, and 8 as well as cumulatively through Years 4, 5, 6, 7, and 8
Time Frame: Years 4, 5, 6, 7, and 8 and cumulatively through Years 4, 5, 6, 7, and 8
Reporting Status: Not Posted

3. Secondary Outcome: Cumulative Pregnancy Percentage
Description: A life table analysis (using Kaplan-Meier) of pregnancies will be performed for the EP population to present the cumulative pregnancy percentage
Time Frame: Years 1 through 3
Population: evaluable for pregnancy population
Measure: Number; unit: Probability
Arm/Group | VeraCept
Number analyzed (Participants) | 1397
Probability
  Year 1 | 0.013
  Year 2 | 0.024
  Year 3 | 0.028

4. Secondary Outcome: Ease of VeraCept Placement
Description: Ease of VeraCept placement will be summarized for the ITT population as reported by the investigator (Very easy, Easy, Neither Easy nor Hard, Hard, Very Hard). (First Attempt)
Time Frame: Visit 1 (Day 1) / VeraCept placement
Population: Number of subjects in ITT population with available information regarding ease of placement at first attempt.
Measure: Count of Participants; unit: Participants
Arm/Group | VeraCept
Number analyzed (Participants) | 1609
Participants
  very easy | 844
  easy | 502
  neither easy nor hard | 160
  hard | 77
  very hard | 26

5. Secondary Outcome: VeraCept Placement Success
Description: The number and percentage of subjects with either a successful or unsuccessful placement will be summarized for the ITT
Time Frame: Visit 1 (Day 1) / VeraCept placement
Measure: Count of Participants; unit: Participants
Arm/Group | VeraCept
Number analyzed (Participants) | 1620
Participants
  successful first attempt of placement | 1549
  successful second attempt of placement | 52
  failed placement | 7
  second attempt not tried | 12

6. Secondary Outcome: Bleeding and Spotting Patterns
Description: Bleeding and spotting patterns will be summarized for the first year of treatment by the number of days in each 28-day cycle with bleeding or spotting, bleeding only, and spotting only
Time Frame: Through year 1
Population: evaluable for cycle control population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VeraCept
Number analyzed (Participants) | 1587
days
  cycle 1: bleeding or spotting: number analyzed (Participants) | 1401
  cycle 1: bleeding or spotting | 11.2 (4.93)
  cycle 1: bleeding only: number analyzed (Participants) | 1401
  cycle 1: bleeding only | 6.4 (3.44)
  cycle 1: spotting only: number analyzed (Participants) | 1401
  cycle 1: spotting only | 4.8 (3.37)
  cycle 2: bleeding or spotting: number analyzed (Participants) | 1271
  cycle 2: bleeding or spotting | 7.8 (3.76)
  cycle 2: bleeding only: number analyzed (Participants) | 1271
  cycle 2: bleeding only | 5.1 (2.57)
  cycle 2: spotting only: number analyzed (Participants) | 1271
  cycle 2: spotting only | 2.7 (2.56)
  cycle 3: bleeding or spotting: number analyzed (Participants) | 1162
  cycle 3: bleeding or spotting | 7.6 (3.73)
  cycle 3: bleeding only: number analyzed (Participants) | 1162
  cycle 3: bleeding only | 5.0 (2.69)
  cycle 3: spotting only: number analyzed (Participants) | 1162
  cycle 3: spotting only | 2.5 (2.43)
  cycle 4: bleeding or spotting: number analyzed (Participants) | 1102
  cycle 4: bleeding or spotting | 7.3 (3.77)
  cycle 4: bleeding only: number analyzed (Participants) | 1102
  cycle 4: bleeding only | 4.9 (2.66)
  cycle 4: spotting only: number analyzed (Participants) | 1102
  cycle 4: spotting only | 2.4 (2.54)
  cycle 5: bleeding or spotting: number analyzed (Participants) | 1036
  cycle 5: bleeding or spotting | 7.2 (3.63)
  cycle 5: bleeding only: number analyzed (Participants) | 1036
  cycle 5: bleeding only | 4.8 (2.60)
  cycle 5: spotting only: number analyzed (Participants) | 1036
  cycle 5: spotting only | 2.4 (2.33)
  cycle 6: bleeding or spotting: number analyzed (Participants) | 946
  cycle 6: bleeding or spotting | 7.0 (3.48)
  cycle 6: bleeding only: number analyzed (Participants) | 946
  cycle 6: bleeding only | 4.8 (2.64)
  cycle 6: spotting only: number analyzed (Participants) | 946
  cycle 6: spotting only | 2.2 (2.27)
  cycle 7: bleeding or spotting: number analyzed (Participants) | 875
  cycle 7: bleeding or spotting | 7.2 (3.79)
  cycle 7: bleeding only: number analyzed (Participants) | 875
  cycle 7: bleeding only | 4.7 (2.73)
  cycle 7: spotting only: number analyzed (Participants) | 875
  cycle 7: spotting only | 2.4 (2.52)
  cycle 8: bleeding or spotting: number analyzed (Participants) | 857
  cycle 8: bleeding or spotting | 7.0 (3.54)
  cycle 8: bleeding only: number analyzed (Participants) | 857
  cycle 8: bleeding only | 4.7 (2.43)
  cycle 8: spotting only: number analyzed (Participants) | 857
  cycle 8: spotting only | 2.3 (2.51)
  cycle 9: bleeding or spotting: number analyzed (Participants) | 797
  cycle 9: bleeding or spotting | 6.9 (3.60)
  cycle 9: bleeding only: number analyzed (Participants) | 797
  cycle 9: bleeding only | 4.6 (2.58)
  cycle 9: spotting only: number analyzed (Participants) | 797
  cycle 9: spotting only | 2.2 (2.36)
  cycle 10: bleeding or spotting: number analyzed (Participants) | 745
  cycle 10: bleeding or spotting | 6.9 (3.40)
  cycle 10: bleeding only: number analyzed (Participants) | 745
  cycle 10: bleeding only | 4.6 (2.44)
  cycle 10: spotting only: number analyzed (Participants) | 745
  cycle 10: spotting only | 2.3 (2.19)
  cycle 11: bleeding or spotting: number analyzed (Participants) | 724
  cycle 11: bleeding or spotting | 6.8 (3.48)
  cycle 11: bleeding only: number analyzed (Participants) | 724
  cycle 11: bleeding only | 4.5 (2.38)
  cycle 11: spotting only: number analyzed (Participants) | 724
  cycle 11: spotting only | 2.2 (2.60)
  cycle 12: bleeding or spotting: number analyzed (Participants) | 703
  cycle 12: bleeding or spotting | 6.8 (3.38)
  cycle 12: bleeding only: number analyzed (Participants) | 703
  cycle 12: bleeding only | 4.7 (2.55)
  cycle 12: spotting only: number analyzed (Participants) | 703
  cycle 12: spotting only | 2.2 (2.24)
  cycle 13: bleeding or spotting: number analyzed (Participants) | 676
  cycle 13: bleeding or spotting | 6.9 (3.50)
  cycle 13: bleeding only: number analyzed (Participants) | 676
  cycle 13: bleeding only | 4.6 (2.50)
  cycle 13: spotting only: number analyzed (Participants) | 676
  cycle 13: spotting only | 2.2 (2.40)

7. Secondary Outcome: Insertion Pain Assessed Immediately After Insertion (First Attempt)
Description: Insertion pain summarized for subjects at first attempt as reported by the subjects
Time Frame: Visit 1 (Day 1), immediately after insertion
Population: Number of subjects in ITT population with available information regarding device placement pain at first attempt.
Measure: Count of Participants; unit: Participants
Arm/Group | VeraCept
Number analyzed (Participants) | 1600
Participants
  no pain | 85
  some pain | 363
  moderately painful | 661
  painful | 406
  very painful | 85

8. Secondary Outcome: Cumulative VeraCept Discontinuation Rates
Description: Cumulative VeraCept discontinuation rates will be summarized using Kaplan-Meier methods for the Safety population.
Time Frame: Years 1 through 3
Population: safety population
Measure: Number; unit: Probability
Arm/Group | VeraCept
Number analyzed (Participants) | 1601
Probability
  Year 1 | 0.195
  Year 2 | 0.329
  Year 3 | 0.419

9. Secondary Outcome: Cumulative VeraCept Expulsion Rates
Description: Cumulative VeraCept expulsion rates will be summarized using Kaplan-Meier methods for the Safety population.
Time Frame: Years 1 through 3
Population: safety population
Measure: Number; unit: Probability
Arm/Group | VeraCept
Number analyzed (Participants) | 1601
Probability
  Year 1 | 0.025
  Year 2 | 0.040
  Year 3 | 0.051

10. Secondary Outcome: Return to Fertility. Only for Subjects Requesting VeraCept Removal to Become Pregnant.
Description: The number and percentage of subjects with each return to fertility response will be summarized for the Safety population.
Time Frame: Subjects will be followed for either 1 year, until they decide to no longer try to conceive or they become pregnant, whichever comes first.
Population: Number of subjects requesting VeraCept removal to become pregnant with known fertility outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | VeraCept
Number analyzed (Participants) | 51
Participants
  pregnancy occurred | 37
  pregnancy did not occur | 14

11. Secondary Outcome: Safety Adverse Events of Special Interest: Pelvic Infection (PID or Endometriosis), Uterine Perforations, and Abdominal Pain
Time Frame: 3 years
Population: safety population
Measure: Number; unit: participants
Arm/Group | VeraCept
Number analyzed (Participants) | 1601
participants
  uterine perforation | 2
  pelvic infection (PID or endometriosis) | 19
  abdominal pain | 111

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- VeraCept: VeraCept™ Intrauterine Contraceptive
  VeraCept: VeraCept Intrauterine Contraceptive is a hormone free, low dose, copper-releasing birth control method
Arm/Group | VeraCept
All-Cause Mortality (participants affected / at risk) | 3/1620
Serious Adverse Events (participants affected / at risk) | 52/1620
Other Adverse Events (participants affected / at risk) | 1551/1601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VeraCept (N=1620)
pyelonephritis (Infections and infestations) | 3 (3)
cellulitis (Infections and infestations) | 2 (2)
pneumonia (Infections and infestations) | 2 (2)
sepsis (Infections and infestations) | 2 (2)
anxiety (Psychiatric disorders) | 2 (2)
depression (Psychiatric disorders) | 2 (2)
suicidal ideation (Psychiatric disorders) | 2 (2)
intentional overdose (Injury, poisoning and procedural complications) | 2 (2)
ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3)
ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
appendicitis (Infections and infestations) | 1 (1)
bacterial colitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
infectious mononucleosis (Infections and infestations) | 1 (1)
pelvic inflammatory disease (Infections and infestations) | 1 (1)
tonsillitis (Infections and infestations) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
drug use disorder (Psychiatric disorders) | 1 (1)
intentional self-injury (Psychiatric disorders) | 1 (1)
psychotic disorder (Psychiatric disorders) | 1 (1)
substance use disorder (Psychiatric disorders) | 1 (1)
substance-induced psychotic disorder (Psychiatric disorders) | 1 (1)
suicide attempt (Psychiatric disorders) | 1 (1)
accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
uterine perforation (Injury, poisoning and procedural complications) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
food poisoning (Gastrointestinal disorders) | 1 (1)
gastric stenosis (Gastrointestinal disorders) | 1 (1)
pancreatitis acute (Gastrointestinal disorders) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 1 (1)
cholecystitis acute (Hepatobiliary disorders) | 1 (1)
cholelithiasis (Hepatobiliary disorders) | 1 (1)
hepatitis (Hepatobiliary disorders) | 1 (1)
hemiparesis (Nervous system disorders) | 1 (1)
migraine (Nervous system disorders) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1)
ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (2)
uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 1 (1)
choledochal cyst (Congenital, familial and genetic disorders) | 1 (1)
chest pain (General disorders) | 1 (1)
anaphylactic reaction (Immune system disorders) | 1 (1)
diabetic complication (Metabolism and nutrition disorders) | 1 (1)
hypoclycaemia (Metabolism and nutrition disorders) | 1 (1)
tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
device breakage (Product Issues) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VeraCept (N=1601)
heavy menstrual bleeding (Reproductive system and breast disorders) | 1246 (3117)
dysmenorrhoea (Reproductive system and breast disorders) | 1172 (2775)
pelvic discomfort (Reproductive system and breast disorders) | 552 (1161)
intermenstrual bleeding (Reproductive system and breast disorders) | 491 (864)
pelvic pain (Reproductive system and breast disorders) | 324 (559)
dyspareunia (Reproductive system and breast disorders) | 128 (160)
vaginal discharge (Reproductive system and breast disorders) | 87 (103)
urinary tract infection (Infections and infestations) | 235 (338)
bacterial vaginosis (Infections and infestations) | 219 (350)
nasopharyngitis (Infections and infestations) | 196 (279)
vulvovaginal mycotic infection (Infections and infestations) | 192 (298)
upper respiratory tract infection (Infections and infestations) | 132 (184)
COVID-19 (Infections and infestations) | 124 (128)
procedural pain (Injury, poisoning and procedural complications) | 292 (317)
post procedural haemorrhage (Injury, poisoning and procedural complications) | 267 (268)
post procedural discomfort (Injury, poisoning and procedural complications) | 97 (98)
nausea (Gastrointestinal disorders) | 123 (168)
headache (Nervous system disorders) | 117 (216)
back pain (Musculoskeletal and connective tissue disorders) | 101 (128)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT03633799/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT03633799/SAP_001.pdf